CLINICAL TRIAL: NCT04016740
Title: Perioperative Multimodal General Anesthesia Focusing on Specific CNS Targets in Patients Undergoing Cardiac Surgeries
Brief Title: The PATHFINDER Study: A Feasibility Trial
Acronym: PATHFINDER
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Associate Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2019P000407
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Delirium
Keywords: Cardiopulmonary Bypass; Cardiac Surgery; analgesics
MeSH Terms: conditions — Coronary Artery Disease; Delirium | interventions — Ropivacaine; Ketamine; Remifentanil; Dexmedetomidine; Rocuronium; Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: 2 roll-in patients followed by 20 patients in the interventional model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal General Anesthesia (Experimental): Intraoperative
  The anesthesiologists involved in this study will be trained to infer differences in anti-nociception, unconsciousness movement and changes during other perioperative events by monitoring EEG. They will also be trained in titrating hypnotic and nociceptic medications based on changes in EEG.
  1. Routine anesthetic induction
  2. Bilateral Pectoro-interfascial block (PIFB) with 20 mL of 0.25% ropivacaine on either side of the sternum after anesthetic induction but before surgical incision
  3. Ketamine (0.06 to 0.12 mg.kg/hr)
  4. Remifentanil (0.05-0.2 mcg/kg/min)
  5. Dexmedetomidine (0.2-1.0 mcg/kg/hr)
  6. Rocuronium intermittent bolus (TOF)
  7. Propofol infusion ± Sevoflurane titrated based on EEG monitoring
  Postoperative
  1. Standard pain management protocol
  2. Dexmedetomidine infusion 0.2-1.4 mcg/kg/hr (EEG guided)
  3. Infusion continued till extubation
  4. Propofol infusion may be added/used for sedation based on the treating physician's discretion
  Interventions: Drug: Ropivacaine; Drug: Ketamine; Drug: Remifentanil; Drug: Dexmedetomidine; Drug: Rocuronium; Drug: Propofol; Drug: Sevoflurane; Device: EEG monitoring
- Standard Practice with EEG monitoring (Other): The initial 2 patients will receive standard anesthesia practice and perioperative EEG monitoring will be recorded to learn the patterns associated with our standard practice.
  Interventions: Device: EEG monitoring

INTERVENTIONS:
Drug: Ropivacaine — Intraoperative bilateral PIFB block with 20 mL of 0.25% Ropivicaine on either side of the sternum after anesthetic induction but before surgical incision
  Arms: Multimodal General Anesthesia
Drug: Ketamine — Intraoperative infusion
  Arms: Multimodal General Anesthesia
Drug: Remifentanil — Intraoperative infusion
  Arms: Multimodal General Anesthesia
Drug: Dexmedetomidine — Intraoperative infusion
  Arms: Multimodal General Anesthesia
Drug: Rocuronium — Intraoperative intermittent bolus
  Arms: Multimodal General Anesthesia
Drug: Propofol — Intraoperative infusion
  Arms: Multimodal General Anesthesia
Drug: Sevoflurane — Intraoperative inhaled as needed
  Arms: Multimodal General Anesthesia
Drug: Dexmedetomidine — Post-operative infusion
  Arms: Multimodal General Anesthesia
Drug: Propofol — Post-operative infusion
  Arms: Multimodal General Anesthesia
Device: EEG monitoring — Perioperative monitoring

SUMMARY:
The main purpose of this study is to determine whether a rational strategy of EEG guided multimodal general anesthesia using target specific sedative and analgesics could result in enhanced recovery after anesthesia and surgery, decrease in postoperative delirium, and decrease in long term postoperative cognitive dysfunction up to 6 months following cardiac surgery.

DETAILED DESCRIPTION:
The main purpose of this study is to determine whether a rational strategy of EEG guided multimodal general anesthesia using target specific sedative and analgesics could result in enhanced recovery after anesthesia and surgery, decrease in postoperative delirium, and decrease in long term postoperative cognitive dysfunction up to 6 months following cardiac surgery.

Specific Aim 1: The feasibility of implementing multimodal general anesthesia strategy in the Operating Rooms (OR) Specific Aim 2: The feasibility of implementing EEG guided sedation until extubation in the Intensive Care Unit (ICU) Specific Aim 3: The enhancement of recovery after surgery (shorter ventilation time, ICU stay, hospital length of stay) Specific Aim 4: To estimate the effect size of decrease in postoperative day (POD) and postoperative cognitive dysfunction (POCD) to power future large randomized trials

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years
2. Undergoing any of the following types of surgery with cardiopulmonary bypass limited to coronary artery bypass surgery (CABG), CABG+valve surgeries and isolated valve surgeries.

Exclusion Criteria:

1. Preoperative left ventricular ejection fraction (LVEF) <30%
2. Emergent surgery
3. Non-English speaking
4. Cognitive impairment as defined by total MoCA score < 10
5. Currently enrolled in another interventional study that could impact the primary outcome, as determined by the PI
6. Significant visual impairment
7. Chronic opioid use for chronic pain conditions with tolerance (total dose of an opioid at or more than 30 mg morphine equivalent for more than one month within the past year)
8. Hypersensitivity to any of the study medications
9. Known history of alcohol (> 2 drinks per day) or drug abuse Active (in the past year) history of alcohol abuse (≥5 drinks/day for men or ≥4 drinks/day for women) as determined by reviewing medical record and history given by the patient
10. Liver dysfunction (liver enzymes > 4 times the baseline, all patients will have a baseline liver function test evaluation), history and examination suggestive of jaundice.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium | Participants will be followed for the duration of the hospital stay, an average of 5 days
  Incidence of delirium will be analyzed in patients treated with the multi-modal approach. Delirium will be defined as an acute change in pre-operative baseline condition with additional features of inattention and either disorganized thinking and altered loss of consciousness, as defined by the Confusion Assessment Method (CAM)Assessment Method (CAM) algorithm postoperatively until discharge.

SECONDARY OUTCOMES:
Time to extubation | Time of ICU admission until time of extubation in ICU, an average of 6 hours
  Time to extubation will be noted from ICU data
Montreal Cognitive Assessment (MoCA) | On the day of discharge, an average of 6 days
  MoCA scores (total possible score is 30 points; a score of 26 or above is considered normal) at discharge will be reported in order to assess the occurrence of postoperative cognitive decline. Study staff trained in administering the assessments will collect the data.
Pain scores | At 4-8 hourly intervals every day until discharge, an average of 6 days
  Patient reported pain scores on a scale from 0-10 (0 no pain,10 extreme pain), until discharge for the index admission.
Total opioid and supplemental analgesic consumption | 48 hours, post-operative
  The total opioid dosage and supplemental analgesic dosage received in the first 48 hours postoperatively will be abstracted from the medical record.
ICU | Time of ICU admission until time of discharge to hospital floor; through the hospital stay, an average of 5 days
  Total duration of stay in ICU for the index admission
ICU/hospital length of stay | Time of stay in the hospital until discharge to floor or rehab, an average of 5 days
  Their stay in the hospital for the index admission
In-hospital complications | 7 days post-op on an average
  stroke, myocardial infarction (MI), acute kidney injury, pneumonia, reintubation, congestive heart failure, sepsis, reopening of sternum and all-cause mortality
Follow up incidence of delirium | Patients will be assessed for delirium at 1 month and 6 months following the date of surgery
  The follow up incidence of delirium will be analyzed at 1 month and 6 months after discharge. Delirium will be defined as an acute change in pre-operative baseline condition with additional features of inattention and either disorganized thinking and altered loss of consciousness, as defined by the MoCA/t-MoCA.

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Brown EN, Pavone KJ, Naranjo M. Multimodal General Anesthesia: Theory and Practice. Anesth Analg. 2018 Nov;127(5):1246-1258. doi: 10.1213/ANE.0000000000003668. PMID 30252709
- [Background] McNicol E, Horowicz-Mehler N, Fisk RA, Bennett K, Gialeli-Goudas M, Chew PW, Lau J, Carr D; Americal Pain Society. Management of opioid side effects in cancer-related and chronic noncancer pain: a systematic review. J Pain. 2003 Jun;4(5):231-56. doi: 10.1016/s1526-5900(03)00556-x. PMID 14622694
- [Background] Volkow ND, Collins FS. The Role of Science in the Opioid Crisis. N Engl J Med. 2017 Nov 2;377(18):1798. doi: 10.1056/NEJMc1711494. No abstract available. PMID 29117474
- [Background] Mulier J. Opioid free general anesthesia: A paradigm shift? Rev Esp Anestesiol Reanim. 2017 Oct;64(8):427-430. doi: 10.1016/j.redar.2017.03.004. Epub 2017 Apr 18. No abstract available. English, Spanish. PMID 28431750
- [Background] MacKenzie KK, Britt-Spells AM, Sands LP, Leung JM. Processed Electroencephalogram Monitoring and Postoperative Delirium: A Systematic Review and Meta-analysis. Anesthesiology. 2018 Sep;129(3):417-427. doi: 10.1097/ALN.0000000000002323. PMID 29912008
- [Background] Depth of anaesthesia monitors - Bispectral Index (BIS), E-Entropy and Narcotrend-Compact M | Guidance and guidelines | NICE [Internet]. [cited 2018 Dec 24];Available from: https://www.nice.org.uk/guidance/dg6
- [Background] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296
- [Background] Wilson PT, Spitzer RL. Major changes in psychiatric nomenclature. Reconciling existing psychiatric medical records with the new American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders. Hosp Community Psychiatry. 1968 Jun;19(6):169-74. No abstract available. PMID 5661463
- [Background] Sauer AM, Slooter AJ, Veldhuijzen DS, van Eijk MM, Devlin JW, van Dijk D. Intraoperative dexamethasone and delirium after cardiac surgery: a randomized clinical trial. Anesth Analg. 2014 Nov;119(5):1046-52. doi: 10.1213/ANE.0000000000000248. PMID 24810262
- [Background] Rudolph JL, Jones RN, Levkoff SE, Rockett C, Inouye SK, Sellke FW, Khuri SF, Lipsitz LA, Ramlawi B, Levitsky S, Marcantonio ER. Derivation and validation of a preoperative prediction rule for delirium after cardiac surgery. Circulation. 2009 Jan 20;119(2):229-36. doi: 10.1161/CIRCULATIONAHA.108.795260. Epub 2008 Dec 31. PMID 19118253
- [Background] Burkhart CS, Dell-Kuster S, Gamberini M, Moeckli A, Grapow M, Filipovic M, Seeberger MD, Monsch AU, Strebel SP, Steiner LA. Modifiable and nonmodifiable risk factors for postoperative delirium after cardiac surgery with cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2010 Aug;24(4):555-9. doi: 10.1053/j.jvca.2010.01.003. Epub 2010 Mar 15. PMID 20227891
- [Background] Arora RC, Djaiani G, Rudolph JL. Detection, Prevention, and Management of Delirium in the Critically Ill Cardiac Patient and Patients Who Undergo Cardiac Procedures. Can J Cardiol. 2017 Jan;33(1):80-87. doi: 10.1016/j.cjca.2016.08.020. Epub 2016 Oct 5. PMID 28024558
- [Background] Delirium: prevention, diagnosis and management | Guidance and guidelines | NICE [Internet]. [cited 2018 Dec 20];Available from: https://www.nice.org.uk/guidance/cg103
- [Background] Pesonen A, Suojaranta-Ylinen R, Hammaren E, Kontinen VK, Raivio P, Tarkkila P, Rosenberg PH. Pregabalin has an opioid-sparing effect in elderly patients after cardiac surgery: a randomized placebo-controlled trial. Br J Anaesth. 2011 Jun;106(6):873-81. doi: 10.1093/bja/aer083. Epub 2011 Apr 6. PMID 21474474
- [Background] Urban MK, Ya Deau JT, Wukovits B, Lipnitsky JY. Ketamine as an adjunct to postoperative pain management in opioid tolerant patients after spinal fusions: a prospective randomized trial. HSS J. 2008 Feb;4(1):62-5. doi: 10.1007/s11420-007-9069-9. Epub 2007 Dec 19. PMID 18751864
- [Background] Ballard C, Jones E, Gauge N, Aarsland D, Nilsen OB, Saxby BK, Lowery D, Corbett A, Wesnes K, Katsaiti E, Arden J, Amoako D, Prophet N, Purushothaman B, Green D. Optimised anaesthesia to reduce post operative cognitive decline (POCD) in older patients undergoing elective surgery, a randomised controlled trial. PLoS One. 2012;7(6):e37410. doi: 10.1371/journal.pone.0037410. Epub 2012 Jun 15. PMID 22719840
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Stoppe C, Fahlenkamp AV, Rex S, Veeck NC, Gozdowsky SC, Schalte G, Autschbach R, Rossaint R, Coburn M. Feasibility and safety of xenon compared with sevoflurane anaesthesia in coronary surgical patients: a randomized controlled pilot study. Br J Anaesth. 2013 Sep;111(3):406-16. doi: 10.1093/bja/aet072. Epub 2013 Apr 11. PMID 23578862
- [Background] Lurati Buse GA, Schumacher P, Seeberger E, Studer W, Schuman RM, Fassl J, Kasper J, Filipovic M, Bolliger D, Seeberger MD. Randomized comparison of sevoflurane versus propofol to reduce perioperative myocardial ischemia in patients undergoing noncardiac surgery. Circulation. 2012 Dec 4;126(23):2696-704. doi: 10.1161/CIRCULATIONAHA.112.126144. Epub 2012 Nov 7. PMID 23136158
- [Background] Papaioannou A, Fraidakis O, Michaloudis D, Balalis C, Askitopoulou H. The impact of the type of anaesthesia on cognitive status and delirium during the first postoperative days in elderly patients. Eur J Anaesthesiol. 2005 Jul;22(7):492-9. doi: 10.1017/s0265021505000840. PMID 16045136
- [Background] Jia Y, Jin G, Guo S, Gu B, Jin Z, Gao X, Li Z. Fast-track surgery decreases the incidence of postoperative delirium and other complications in elderly patients with colorectal carcinoma. Langenbecks Arch Surg. 2014 Jan;399(1):77-84. doi: 10.1007/s00423-013-1151-9. Epub 2013 Dec 13. PMID 24337734
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Derived] Shanker A, Abel JH, Narayanan S, Mathur P, Work E, Schamberg G, Sharkey A, Bose R, Rangasamy V, Senthilnathan V, Brown EN, Subramaniam B. Perioperative Multimodal General Anesthesia Focusing on Specific CNS Targets in Patients Undergoing Cardiac Surgeries: The Pathfinder Feasibility Trial. Front Med (Lausanne). 2021 Oct 14;8:719512. doi: 10.3389/fmed.2021.719512. eCollection 2021. PMID 34722563